CLINICAL TRIAL: NCT00377533
Title: Wheelchair Handling Skills of Caregivers: Comparison Between Conventional Rear Anti-tip Devices and a New Design
Brief Title: Wheelchair Handling Skills of Caregivers: Comparison Between Anti-tip Devices and a New Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDHA013
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2010-04-05 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
Keywords: wheelchairs; caregivers; skills

INTERVENTIONS:
Device: wheelchair rear anti-tip device — assistive device

SUMMARY:
Currently available wheelchairs are often fitted with conventional rear anti-tip devices (C-RADs) to prevent wheelchair rear tips. The limitations of C-RADs have provided an incentive for the design of rear anti-tip devices that permit more rear tip without compromising safety (Arc-RADs).

The purpose of this study is to test the hypothesis that caregivers handling occupied wheelchairs equipped with Arc-RADs have higher success rates on RAD-relevant skills than caregivers handling wheelchairs equipped with C-RADs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* alert, able and willing to follow instructions
* wheelchair users: patients at the Nova Scotia Rehabilitation Centre
* wheelchair users:permission of physician to participate in the study
* caregiver:must provide at least part-time wheelchair-handling care for the wheelchair user in this study, a minimum of one hour per week on average

Exclusion Criteria:

* wheelchair users:suffer from any unstable medical, emotional, or physiological conditions that may interfere with participation
* caregivers:medical condition of their upper limbs, heart or lungs that might cause them discomfort or endanger them when pushing or pulling an occupied wheelchair

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Wheelchair Skills Test | day

CONTACTS AND LOCATIONS:
Overall Officials: Lee Kirby, MD, FRCPC, Principal Investigator — Dalhousie University, QEII Health Sciences Centre
Locations (1):
- QEII Health Science Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- See also: Wheelchair skills program — http://www.wheelchairskillsprogram.ca/